CLINICAL TRIAL: NCT06759961
Title: Post-transplant Thrombotic Microangiopathy: Evaluation of Outcomes at the Bologna Kidney Transplant Centre
Acronym: PT-TMA2022
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PT-TMA2022
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Microangiopathy; Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a retrospective-prospective, single-centre, non-pharmacological, retrospective tissue study carried out for scientific and health protection purposes. It involves the systematic collection of clinical information from patients diagnosed with PT-TMA

DETAILED DESCRIPTION:
The primary objective is to calculate the incidence of PT-TMA in a large cohort of kidney transplant patients and to assess the association between PT-TMA and renal transplant outcome.

It provides for the systematic collection of clinical information of patients with a diagnosis of PT-TMA, starting from 01/06/2016 until the approval of the study by the Ethics Committee and the issuance of the authorisation by the Director General of the IRCCS; the evaluation of the prospective data will be carried out starting from the approval of the study by the Ethics Committee and the issuance of the authorisation by the Director General of the IRCCS and will continue for 10 years. Patients enrolled prospectively will be treated according to clinical practice, in accordance with the judgement of the Physician

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Living kidney transplant recipient, brain death cadaver donor, cardiac death cadaver donor, single kidney transplant, double kidney transplant, combined kidney transplant
* Acquisition of Informed Consent to participate in the study and to process personal, special and genetic data

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the period from 01/06/2016 until 01/09/2022 at the Transplant Centre of the Nephrology, Dialysis, Transplantation Unit of our hospital, 715 kidney transplants were performed. The incidence of post-transplant thrombotic microangiopathy varies according to literature data up to a maximum of 14-15%. The estimated population size as the object of the retrospective study is therefore approximately 750 patients in total and approximately 100 patients with PT-TMA. The size of the population as the subject of the prospective study is approximately 1200 transplanted patients with approximately 150/180 patients developing PT-TMA.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PT-TMA and renal graft outcome | 15 days, 1 month, 6 months after transplantation and then every 6 months thereafter
  * The incidence of PT-TMA will be assessed in this cohort by considering the number of events over the total number of patients in the observation period.
  * The renal graft outcome will be assessed by considering graft failure events (return to ESKD, kidney retransplantation) and calculating the eGFR at 15 days, 1 month, 6 months after transplantation and then every 6 months thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Comai, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Sant'Orsola University Hospital - Nephrology, Dialysis and Transplant Unit, Bologna, BO, Italy